CLINICAL TRIAL: NCT07216638
Title: Pediatric Behavioral Health Integrated Care: Indiana Statewide Strategic Plan to Address the Growing Mental Health Crisis
Acronym: PEDS-IBH
Status: Enrolling by invitation | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Matthew Aalsma, Johnathan & Jennifer Simmons Professor of Pediatrics & Director of the Child Health Services Research Division and the Adolescent Behavioral Health Research Program, Indiana University
Other Study IDs: 20891; 0069660 (Other Grant/Funding Number: Indiana Family and Social Services Administration, Division of Mental Health and Addiction)
Record Dates: First submitted 2025-09-23; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Implementation Research; Depressive Disorder; ANXIETY DISORDERS (or Anxiety and Phobic Neuroses); Conduct Disorders in Children; Pediatric Mental Health Services
Keywords: Implementation; Pediatric Mental Health Services; Pediatric Mental Health; Depression; Anxiety; Conduct Disorders
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Phobic Disorders; Depression; Conduct Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Care Practice As Usual: Data are collected regarding standard primary care practice and outcomes before the implementation of PEDS-IBH
- Integrated Behavioral Health with PEDS-IBH Resources: Participating clinics receive a system-level intervention, PEDS-IBH. Designed to improve youth mental health detection and treatment.

SUMMARY:
This research is designed to analyze the implementation and fidelity of Pediatric Integrated Behavioral Health (PEDS-IBH). PEDS-IBH is a multifaceted project designed to address the pediatric mental health crisis by providing prompt and continuing mental health resources to pediatric patients in the primary care setting. The belief is the best way to combat this crisis is through early detection and treatment. Primary care providers (PCP) play a vital role in helping youth with mental health disorders because most youth see their PCP on a yearly basis for their annual well-child visits. However, PCPs have many barriers to treating their young patients with mental health disorders: lack of training, resources, and support to deliver interventions, limited time with patients, and the only available referral options often come with long wait times for an appointment or are at a distance to far for the patient to travel.

Indiana University Health (IU Health) has sought to address these concerns by implementing the PEDS-IBH program in 25 different pediatric primary care sites throughout the state of Indiana. Each location will focus on early detection through screening and will have an assigned social worker with either a bachelors or master's level degree. Social workers will administer FIRST or MATCH therapy respectively to those who have been referred and meet the qualifications within the patient's "home" IU Health Clinic. The goal of this project is to learn if clinics participating in PEDS-IBH will increase in early detection and delivery of effective youth mental health treatment. Ultimately leading to better health outcomes when compared to standard primary care detection and treatment.

The research portion of PEDS-IBH has three aims, (Aim 1) Evaluate the implementation of the Peds IBH program including the uptake/adoption of and fidelity to the program. (Aim 2) Explore the facilitators and barriers to the implementation of the Peds IBH program. (Aim 3) Compare youth connection to behavioral health care pre- and post-implementation of the Peds IBH program, including time from referral to engagement in behavioral health services and use of emergency department, inpatient, and residential placements. The research team will interview and survey willing PCP's, clinic managers, and other clinic staff to gather information to address the aforementioned aims.

DETAILED DESCRIPTION:
The mental health crisis in the United States and in Indiana is growing at a rapid and alarming pace. Indiana ranks 43rd in behavioral health workforce availability and 23rd in youth prevalence of mental illness. With suicide being the 2nd leading cause of death among children ages 10-14 in Indiana and the growing rate of substance use and abuse, this project is focused on addressing mental health issues before the issues reach crisis levels.

The PEDS-IBH project is a comprehensive initiative aimed at addressing the growing mental health needs of pediatric patients by integrating timely and ongoing behavioral health support directly into primary care. Providers can refer children to the program when mental health, behavioral, or substance use concerns are identified-whether raised by the patient or caregiver, observed by the provider, or uncovered through routine screening. A key component of the program is universal mental health screening, which helps normalize behavioral health care as part of overall wellness. Clinics involved in the PEDS-IBH initiative use the K-CAT (Kiddie Computer Adaptive Test), a validated, adaptive screening tool for children ages 7 to 17, to assess a range of mental health issues, including depression, anxiety, ADHD, conduct disorders, and suicidality, based on both self and caregiver reports.

When concerns are identified, children can be referred to virtual Riley therapy groups or in-clinic behavioral health providers trained to deliver evidence-based treatments like FIRST or MATCH, depending on their professional training level. FIRST is a structured, short-term intervention validated for children as young as five, focused on treating mild to moderate mental health symptoms by teaching key cognitive-behavioral skills. The program is designed to intervene early and efficiently, while also ensuring that children with more complex or severe concerns-such as suicidality or significant developmental conditions-are connected to appropriate higher-level specialty care. Through this model, PEDS-IBH enhances the pediatric medical home by supporting early identification, timely intervention, and coordinated mental health treatment.

By analyzing a multifaceted intervention designed to help change the cultural and procedural norms of the pediatric primary care setting regarding pediatric mental health treatment. This study looks to ensure the workforce in primary care clinics are equipped to detect and treat mental health disorders in a timely and convenient manner for their patients.

Pediatric primary care providers (PCPs) are well-positioned to play a vital role in managing adolescent mental health needs, as most youth attend annual well-child visits and PCPs are already engaged in treating mental health conditions. However, systemic barriers within primary care limit their ability to expand access to necessary behavioral health services. Many PCPs struggle to conduct adequate screening or assessment due to time constraints during appointments, making it difficult to implement even brief mental health interventions. Furthermore, while treatments and specialists may exist, workforce shortages in community-based behavioral healthcare often leave PCPs without viable referral options, compounding the challenge.

In addition to limited resources and training, PCPs may feel unqualified to independently address more complex mental health conditions, which can lead to uncertainty in how best to support affected adolescents. These challenges are exacerbated by persistent stigma within primary care settings, where providers and staff may hold negative attitudes toward individuals with behavioral health conditions, reducing their willingness to engage in necessary care. To overcome these barriers, empirically supported, team-based models are needed to shift norms within primary care, reduce stigma, and strengthen the behavioral health workforce to meet the evolving needs of adolescents.

ELIGIBILITY:
Inclusion Criteria: For providers and staff recruited to complete surveys, focus groups, and/or interviews:

1. member of participating pediatric primary care team in participating PEDS-IBH clinics
2. at least 18 years old
3. speaks and understanding English.

Inclusion Criteria for administrative data:

1. patient at one of the participating pediatric primary care team
2. 5-18 years old -

Exclusion Criteria:

* N/A

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IU Health and Riley Primary Care Clinics
Sampling Method: Non-Probability Sample
Enrollment: 575 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Physician Belief Scale | Surveys will be collected prior to implementation, then continue every six months for a total of 2 years.
  Attitudinal constructs will be measured using a 14-item measure indexing providers attitudes toward management of psychosocial problems and comprises of two subscales (Belief and Feeling, Burden) (McLennan et al., 1999). Including one item to asses burnout. Utilizes a 5 point Likert Scale, with 1 being Strongly Disagree and 5 Being Strongly Agree.
Organizational Constructs | Surveys will be collected prior to implementation, then continue every six months for a total of 2 years.
  Implementation Climate Scale, an 18-item measure of the degree to which the organizational climate is supportive of evidence-based practice (EBP) adoption and consists of six subscales (focus on EBP, educational support for EBP, recognition for EBP, rewards for EBP, selection for EBP, and selection for openness). Utilizes a 5 point Likert-type Scale, with 0 being "Not at All" and 4 being "Very great extent". Implementation Leadership Scale (Aarons et al., 2014), a 6-item measure of leadership support for EBP, specifically Peds IBH, implementation and Primary Care Dynamics Survey. Which is also a 5 point Likert-type Scale, with 0 being "Not at All" and 4 being "Very great extent". And an 11-item measure of primary care team dynamics (Song et al., 2015), from which we included two subscales (process for communication and information exchange, and acting and feeling like a team). Which uses a Utilizes a 5 point Likert Scale, with 1 being "Strongly Disagree" and 5 being "Strongly Agree".
Implementation Outcomes | Surveys will be collected prior to implementation, then continue every six months for a total of 2 year.
  Behavioral Health Screening, Referral, and Consultation Experience and Implementation, developed to assess provider-reported behavior and includes seven items at pre-implementation and 10 at mid- and post-implementation. All questions using a visual analogue scale, with 0 being the lowest and 100 being the highest.
Acceptability, Feasibility, and Appropriateness Measure | Surveys will be collected prior to implementation, then continue every six months for a total of 2 year.
  Acceptability of Intervention, Intervention Appropriateness, and Feasibility of Intervention Measure, a 12-item measure of the acceptability, feasibility, and appropriateness of the implemented program, Peds IBH. Which uses a Utilizes a 5 point Likert Scale, with 1 being "Completely Disagree" and 5 being "Completely Agree".
System Usability Scale | Surveys will be collected prior to implementation, then continue every six months for a total of 2 year.
  Systems Usability Scale, a 12-item measure of the usability and learnability of a given system, which was adapted to assess the Kiddie-Computerized Adaptive Tests (K-CAT) screening tool. Utilizes a 5 point Likert Scale, with 1 being Strongly Disagree and 5 Being Strongly Agree.
Provider Report of Sustainment Scale | Surveys will be collected prior to implementation, then continue every six months for a total of 2 years.
  Provider Report of Sustainment Scale, a 3-item measure of the sustainability or continued use of the implemented program, Peds IBH. Utilizes 5 point Likert Scale, with the lowest point being "Not at all" and the highest point being "To a Very Great Extent".
Confidence in Ability to Identify Behavioral Health Concerns and Connect to Services | Surveys will be collected prior to implementation, then continue every six months for a total of 2 years.
  Barriers encountered when implementing the Peds IBH program, and suggested improvement/resources/trainings using seven items. Utilizing an 11 point Likert Scale, with O being the lowest and 10 being the highest. As well as 3 open-ended text box questions.
Screening Rates | From clinical trial launch, data will be collected twice a year, for a total of four years
  Percent of youth screened for Mental Health Disorders. Measuring screening rates as the percent of 7- to 17-year-olds who have PSC-17 and/or PHQ-2/-9 screening results.
Referral Rates | From clinical trial launch, data will be collected twice a year, for a total of four years.
  Percent of youth referred to FIRST therapy for treatment. Referral rates to the Peds IBH program as the percent of patients with a positive screen who are referred to the Peds IBH program.
PEDS-IBH Implementation Opinion via Clinic Interviews | Interviews will be collected prior to implementation, then continue every six months for a total of 1 year
  Semi-structured interviews involving a Nurse/MA, PCP, and clinic manager of participating PEDS-IBH clinics. Interviews will be conducted virtually by a member of the implementation team. Interviews will inquire about the process for determining if a youth is in need of behavioral health services and shifts in this process following Peds IBH program implementation; their clinic's behavioral health screening and referral process; and Peds IBH program feasibility, fit, integration, implementation, and barriers and facilitators to implementation.
Provider 2 Provider (P2P) Consultation Calls | From clinical trial launch, data will be collected twice a year, for a total of four years.
  Number of P2P Consultation Calls. Data will be provided from the BeHappy and AAA consultation lines on number of consultation calls from participating clinics.
Top Problem Assessment | From clinical trial launch, data will be collected twice a year, for a total of four years.
  Youth and their caregiver(s) who participate in the FIRST intervention will complete the Kiddie-Computerized Adaptive Tests (K-CAT) at pre- and post-treatment and Top Problems Assessment at each session to evaluate treatment outcomes. The K-CAT and Top Problems Assessment will be administered as part of routine care for youth receiving the FIRST intervention. The Top Problems Assessment is an idiographic assessment of youth and caregiver identified top problems.
Assess Youth Engagement in Services | From clinical trial launch, data will be collected twice a year, for a total of four years.
  Measure rates of youth engagement in the Peds IBH program. This data will be collected through administrative data in the EHR. We will measure 1) the percent of youth referred to the Peds IBH program who schedule a Peds IBH assessment appointment, 2) the percent of youth who have a scheduled assessment appointment who attend the appointment, 3) the percent of youth indicated as appropriate for Peds IBH services who attend at least one session of FIRST, and 4) the number of total FIRST sessions attended.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Hulvershorn, MD, Principal Investigator — Indiana University/Indiana University Health; Matthew C Aalsma, PhD, Principal Investigator — Indiana University/Indiana University Health
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States